CLINICAL TRIAL: NCT03396419
Title: A Sub-Study of the ImpACT-24B Trial (CLP1000500) Assessing Brain Collateral Blood Flow Enhancement Following Spheno-Palatine Ganglion (SPG) Stimulation in Subjects With Acute Ischemic Stroke
Brief Title: IMPACT- 24col Collateral Blood Flow Assessment Following SPG Stimulation in Acute Ischemic Stroke (ImpACT-24B Sub-Study)
Status: Terminated | Type: Observational
Why Stopped: Terminated following the completion of ImpACT-24B study
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP1050611
Record Dates: First submitted 2017-09-27; First posted 2018-01-11 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Isch. Stk pts treat. w/SPG stimul.: Following implantation (according to the ImpACT-24B protocol), subjects will be transferred to the angio suite. A baseline brain digital subtraction angiography (DSA) will then be performed by a trained physician prior to initiation of SPG stimulation according to the ImpACT-24B protocol.
  Following the first SPG stimulation cycle of 4 minutes, a post-stimulation DSA will be performed.
  Based on the results of the post-stimulation DSA, the physician may perform an additional DSA following the second SPG stimulation cycle.
  The subject will then be transferred to the stroke department and will continue treatment according the ImpACT-24B protocol.

SUMMARY:
The purpose of the ImpACT-24col sub-study is to explore effect of SPG stimulation on the augmentation of collateral blood flow and to relate it to the subject's cerebral blood flow status, the extent of the collateral vessel potency prior to the stimulation and the relation of the vessel occlusion site to the vasodilatory effect by using digital subtraction angiography (DSA), the gold standard imaging technique to demonstrate collateral blood flow dynamics. The results of this study will further promote the knowledge towards optimization of SPG stimulation to treat acute ischemic stroke patients.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability, death and health care expenditure. It is the second most common cause of death worldwide, exceeded only by heart disease. Ischemic stroke constitutes 83 to 90% of stroke cases in western countries. Occlusion of the Middle Cerebral Artery (MCA) in the anterior circulation, or its branches is the most common site, accounting for approximately 90% of infarcts and two thirds of all first strokes. Available therapies include intravenous recombinant tissue plasminogen activator (IV rt-PA) and mechanical recanalization using thrombectomy (MT) devices. Both treatment approaches are primarily focused on recanalization, i.e. aiming to restore artery potency and brain perfusion to reduce the volume of cerebral infarction which thereby reduces functional deficits. Recent meta-analysis of the results demonstrated that although MT is an effective therapy, still over 50% of the treated patient do not recover. IV rt-PA treatment suffers from similar, more significant, lack of effect in majority of patients. This lack of treatment success is probably a result of inadequate micro circulatory collateral blood flow in the involved brain tissue. Treatment targeting collateral cerebral blood flow augmentation is a promising therapy, either as a stand-alone treatment, or as a complementary treatment post recanalization. BrainsGate's device, the ISS, augments brain perfusion through the collateral circulation. The augmentation of collateral blood flow is a result of stimulation of the Spheno-Palatine Ganglion (SPG). The SPG is the source of parasympathetic innervations to the anterior cerebral circulation, which comprises the middle cerebral artery, the anterior cerebral artery, and their tributaries. Studies in rodents, dogs and monkeys have demonstrated that stimulation of SPG neurons leads to a profound ipsilateral increase in the CBF because of arterial vasodilatation, and that this leads in turn to augmentation of tissue perfusion (see Figure 1). Moreover, previous studies, including histopathologic studies in humans have revealed that the main neurotransmitters of this neuronal pathway are acetylcholine (ACh), vasoactive intestinal peptide (VIP), and nitric oxide (NO). It is interesting to note that NO is best known for its potent vasodilatory activity and its capacity for neuroprotection and neurogenesis. Several studies have demonstrated that the cerebral vasodilatation induced by SPG stimulation is indeed mediated through NO mechanisms and that ablation of the SPG efferents to the cerebral vasculature leads to an increased infract size in MCA-occluded rats. So far, imaging studies aiming to demonstrate collateral blood flow augmentation due to SPG stimulation were not yet performed in human stroke patients. It is highly important to study the effect of SPG stimulation on the augmentation of collateral blood flow and to relate it to the subject's cerebral blood flow status, the extent of the collateral vessel potency prior to the stimulation and the relation of the vessel occlusion site to the vasodilatory effect. The purpose of the ImpACT-24col sub-study is to explore these important questions by using digital subtraction angiography (DSA), the gold standard imaging technique to demonstrate collateral blood flow dynamics. The results of this study will further promote the knowledge towards optimization of SPG stimulation to treat acute ischemic stroke patients. The ImpACT-24col study will be a sub-study of the ImpACT-24B trial and eligible patients will be enrolled to both trials.

ELIGIBILITY:
The Inclusion/Exclusion criteria are those of the ImpACT-24B trial (CLP1000500).

Additionally, subjects will be excluded from the ImpACT-24col sub-study if DSA is contraindicated (such as allergy to the contract media, etc.).

Inclusion Criteria:

1. Age: Between 40 years and 80 years for male and 85 for female subjects
2. Clinical diagnosis of an acute ischemic stroke in the Carotid, Middle or Anterior Cerebral Artery territories
3. Imaging findings demonstrating signs of ischemia in the anterior circulation, consistent with the clinical diagnosis
4. Baseline NIHSS ≥ 7 and ≤ 18 within 2 hours prior to implantation.
5. Ability to initiate treatment within 8- 24 hours from stroke onset
6. Signed informed consent from patient him/herself or legally authorized representative if applicable

Exclusion Criteria:

1. Intracranial hemorrhage or hemorrhagic transformation
2. Massive stroke
3. Acute ischemic stroke in the posterior circulation
4. Minor stroke
5. Treated with IV-tPA ,IA-tPA or neurothrombectomy devices for the current stroke
6. Previous stroke in the last 6 months or pre-existing disability
7. Patients with bleeding propensity or any condition in the oral cavity that prevents implantation
8. Clinical signs and symptoms or imaging evidence of bilateral stroke.
9. Treated with IV-tPA ,IA-tPA or neurothrombectomy devices for the current stroke.
10. Known cerebral arteriovenous malformation, cerebral aneurysm.
11. Clinical suspicion of septic embolus.
12. Uncontrolled hypertension (systolic >185 mmHg and/or diastolic >110 mmHg)
13. Serious systemic infection.
14. Women known to be pregnant or having a positive or indeterminate pregnancy test.
15. Patients with other implanted neural stimulator/ electronic devices (pacemakers).
16. Life expectancy < 1 year from causes other than stroke.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Acute Ischemic Stroke in the anterior circulation enrolled to the ImpACT-24B study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Collateral blood flow grades difference following SPG stimulation. | Day 1
  The difference between the collateral blood flow grades, assessed by DSA, at baseline and following SPG stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Slolberg, Dr., Study Director — BrainsGate
Locations (1):
- High Technology Medical Center University Clinic LTD., Tbilisi, Georgia